CLINICAL TRIAL: NCT03926091
Title: A Prospective, Multisite, Randomized, Open-label Phase III Clinical Trial (CLOVER Study)Comparing 4 Cycles With 6 Cycles of TC (Docetaxel+Cyclophosphamide) Adjuvant Chemotherapy for 1-3 Lymph Node Positive ER+/HER2- Early Breast Cancer
Brief Title: Study Comparing 4 Cycles With 6 Cycles of TC (Docetaxel+Cyclophosphamide) Adjuvant Chemotherapy for 1-3 Lymph Node Positive ER+/HER2- Early Breast Cancer
Acronym: CLOVER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOVER
Record Dates: First submitted 2019-03-31; First posted 2019-04-24 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: docetaxel; cyclophosphamide; adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Arm 1：6 cycles of TC (Docetaxel 75 mg/m^2 ivgtt d1+Cyclophosphamide 600 mg/m^2 iv d1, 21 days per cycle).
  Arm 2：4 cycles of TC (Docetaxel 75 mg/m^2 ivgtt d1+Cyclophosphamide 600 mg/m^2 iv d1, 21 days per cycle).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 cycles of TC adjuvant chemotherapy (Experimental): 4 cycles of TC (Docetaxel 75 mg/m^2 ivgtt d1+Cyclophosphamide 600 mg/m^2 iv d1, 21 days per cycle).
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide
- 6 cycles of TC adjuvant chemotherapy (Active Comparator): 6 cycles of TC (Docetaxel 75 mg/m^2 ivgtt d1+Cyclophosphamide 600 mg/m^2 iv d1, 21 days per cycle).
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel — Docetaxel chemotherapy (injection)
  Other Names: docetaxel injection
Drug: Cyclophosphamide — Cyclophosphamide chemotherapy (injection)
  Other Names: Cyclophosphamide injection

SUMMARY:
This is a prospective, multisite, randomized, open-label Phase III clinical trial (CLOVER study) comparing 4 cycles with 6 cycles of TC (docetaxel+cyclophosphamide) adjuvant chemotherapy for 1-3 positive lymph node, ER+/HER2- early breast cancer patients.

DETAILED DESCRIPTION:
While TC (docetaxel+cyclophosphamide) adjuvant chemotherapy is one of the preferred regimens for early breast cancer, we have yet to determine the optimum number of cycles for TC adjuvant chemotherapy. In this prospective, open-label clinical trial, estrogen receptor (ER)-positive, human epidermal growth factor receptor 2 (HER2)-negative early breast cancer patients with 1-3 positive lymph nodes will be randomized into either 4 cycles or 6 cycles of TC adjuvant chemotherapy. The safety and efficacy of each group will be assessed through disease-free survival (DFS), invasive disease free survival (iDFS), distant disease free survival (DDFS), overall survival (OS) and adverse effects (AE) as graded by Common Terminology Criteria for Adverse Events (CTCAE) 4.0.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-70 years old;
2. Patient has localized invasive breast carcinoma with1-3 positive lymph nodes, and is ER+/HER2- confirmed by histopathology after early breast cancer surgery（HER2-negative breast cancer (based on most recently analyzed biopsy) defined as a negative in situ hybridization test or an Immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (Fluorescence in situ hybridization (FISH), Chromogenic in situ hybridization (CISH) , or Silver in situ hybridization (SISH)) test is required by local laboratory testing.), with at least one of the following conditions: (1) histological grade III; (2) Ki67 ≥ 30%; (3) progesterone receptor (PR) ≤ 20% positive; (4) age less than 35 years; (5) extensive vascular tumor thrombus; (6) multigene detection recurrence score (RS) >25;
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN，and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula).
5. Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

1. Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy）;
2. Has bilateral breast cancer;
3. Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
4. Has metastatic (Stage 4) breast cancer;
5. Has any >T4 lesion (UICC1987) (with skin involvement, mass adhesion and fixation, and inflammatory breast cancer);
6. Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
7. Patients participating in other clinical trials at the same time;
8. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
9. Has known allergy to taxane and excipients.
10. Has severe or uncontrolled infection;
11. Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders;
12. the researchers judged patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2172 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Invasive disease free survival | 5 year

SECONDARY OUTCOMES:
disease free survival | 5 years
distant disease free survival | 5 years
overall survival | 5 years
adverse effects | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD, PhD, Principal Investigator — Fudan University
Locations (14):
- China (14):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yet-Sen Memorial Hospital, Sun Yet-Sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Bethune Hospital of Jilin University (The First Hospital of Jilin University), Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - OB/GYN Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, ZheJiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou, Zhejiang